CLINICAL TRIAL: NCT00513266
Title: Oxaliplatin-CPT-11-5-FU-Leucovarin + Bevacizumab and Cetuximab (OCFL-BC) as a Combination Regimen for Systemic Treatment of Advanced Colorectal Carcinoma With Potentially Resectable Liver and/or Lung Metastases. A Phase II Study
Brief Title: Combination Chemotherapy and Monoclonal Antibody Therapy in Treating Patients With Advanced Colorectal Cancer With Liver Metastases or Lung Metastases That Are Potentially Removable by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000559146; CHUV-CH-OCFL-BC; EU-20741
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-06

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: recurrent rectal cancer; stage IV rectal cancer; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases; lung metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Cetuximab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant; Biopsy; Neoadjuvant Therapy

INTERVENTIONS:
Biological: bevacizumab
Biological: cetuximab
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: biopsy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, irinotecan, fluorouracil and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab and cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy together with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with monoclonal antibody therapy works in treating patients with advanced colorectal cancer with liver metastases or lung metastases that are potentially removable by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the pathological complete response (CR) rate in resected patients assessed on lesions of less than or equal to 30 mm in size.

Secondary

* To determine the clinical CR rate in all patients.
* To determine toxicity and tolerability of this regimen (pre- and postoperative toxicity).
* To evaluate perioperative safety in these patients.
* To determine disease-free survival (time to progression in unresected patients) and overall survival of the whole study population.
* To determine resectability in these patients.
* To evaluate markers that predict the occurrence of a pathological CR or a non-response in pathological material (resected liver metastasis) and biological material collected from these patients.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, and 29, oxaliplatin IV over 2 hours on days 1 and 15, irinotecan hydrochloride IV over 30 minutes on days 8 and 22, fluorouracil IV over 24 hours on days 1, 8, 15, and 22, leucovorin calcium IV on days 1, 8, 15, and 22, and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 5 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients who are able to undergo liver resection receive bevacizumab on day 1 only of course 3 and undergo liver resection 3 weeks after chemotherapy. Beginning 4 weeks after liver resection, patients receive 2 additional courses of chemotherapy as adjuvant therapy.

Patients undergo tumor tissue and blood sample collection periodically for biological studies. Samples are analyzed for markers that predict the occurrence of a complete pathological response (pCR) or a non-response.

After completion of study treatment, patients are followed every 3 months for the first 2 years and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma
* Bidimensionally measurable metastatic disease limited to the liver and considered curatively resectable after response to systemic therapy as assessed by a surgical board

  * Additional metastatic disease to the lungs consisting of no more than 3 potentially resectable lesions allowed
  * Must have at least one lesion of 30 mm or less

Exclusion criteria:

* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., uncontrolled seizure with standard medical therapy or history of stroke)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Performance status ≤ 1
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine 1.25 x upper limit of normal (ULN)
* Bilirubin 1.25 x ULN (1.5 x ULN if liver metastasis)
* AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastasis)
* Woman and men of childbearing age must use adequate contraception

Exclusion criteria:

* Pregnancy (positive serum pregnancy test) or lactation
* Chronic diarrhea ≥ grade 2
* Other serious illness or medical condition including any of the following:

  * Unstable cardiac disease requiring treatment
  * Congestive heart failure or angina pectoris even if medically controlled
  * Significant arrhythmias
  * History of significant neurologic or psychiatric disorders including psychotic disorders, dementia, or seizures that would prohibit the understanding and giving of informed consent
  * Active uncontrolled infection
  * Severe hypercalcemia
  * Other serious underlying medical condition that could impair the ability of the patient to participate in the study
  * Neuropathy > grade 1 of any etiology
* Known DPD deficiency
* Known severe polyneuropathy
* Known allergy to Chinese hamster ovary cell proteins, other recombinant human or humanized antibodies, any excipients of bevacizumab formulation, or any other study drugs
* Chronic inflammatory bowel disease
* Acute or subacute intestinal occlusion
* History of previous arterial thromboembolism
* Uncontrolled hypertension
* Evidence of bleeding diathesis or coagulopathy
* Serious nonhealing wound, ulcer, or bone fracture
* History of tumor other than basocellular carcinoma of the skin
* Peripheral neuropathy > grade 1 of any origin (e.g., alcohol)
* Significant traumatic injury within 28 days prior to study treatment

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* No prior chemotherapy for metastatic disease

  * Prior adjuvant chemotherapy permitted if interval since last treatment administration and recurrence is > 6 months
* Major surgical procedure or open biopsy within 28 days prior to study treatment or anticipation of the need for major surgical procedure during the course of the study
* Treatment in a clinical trial within 30 days prior to study entry
* Concurrent treatment with other experimental drugs or other anticancer therapy
* Current or recent use (within 10 days prior to study treatment) of full-dose oral or parenteral anticoagulants for therapeutic purposes
* Chronic daily treatment with aspirin (> 325 mg/day)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Pathological complete response rate of lesions of less than or equal to 30 mm in size assessed by pathologic examination in resected specimens

SECONDARY OUTCOMES:
Response as assessed by NCIC criteria
Toxicity as assessed by NCIC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Roth, MD, Study Chair — Hopital Cantonal Universitaire de Geneve
Locations (4):
- Switzerland (4):
  - Kantonspital Aarau, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Hopital Regional de Sion-Herens-Conthey, Sion